CLINICAL TRIAL: NCT02074423
Title: A Randomized, Controlled, Double-blind, Cross-over Clinical Trial, Evaluating the Effect of MealShape™ on the Postprandial Glycemia After Eating Standard Food, in Healthy Volunteers.
Brief Title: A Human Clinical Trial Evaluating the Effect of MealShape™ on Blood Glucose Level Following Consumption of Standard Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dialpha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-026
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Postprandial Glycemia; Postprandial Insulinemia
Keywords: Cinnamon extract; Postprandial glycemia; Glycemic index; Pre-diabetes; Metabolic syndrome
MeSH Terms: conditions — Glucose Intolerance; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MealShape cinnamon extract (Experimental): Intake of 2 capsules of 500 mg MealShape 30 minutes before consumption of a standard meal (white bread)
  Interventions: Dietary Supplement: MealShape cinnamon extract
- Placebo (Placebo Comparator): Intake of 2 capsules of 500 mg placebo, composed of 20% microcrystalline cellulose and 80% dicalcium phosphate, 30 minutes before consumption of a standard meal (white bread)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MealShape cinnamon extract — Acute administration of 1 g PO (2 capsules of 500 mg)
  Arms: MealShape cinnamon extract
Dietary Supplement: Placebo — Acute administration of 1 g PO (2 capsules of 500 mg)
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect of MealShape, a Ceylon cinnamon extract (Cinnamomum zeylanicum) on blood glucose and insulin response after consumption of a standard meal composed of white bread, in healthy male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, able to read and write, aged from 18 to 45 years inclusive at time of screening
* Good physical condition
* Body Mass Index (BMI) ≥ 18,5 and < 25 kg/m²
* Written informed consent provided prior to screening, after receiving and understanding the subject information
* Stable body weight (< 5% variation) within the last 3 months prior to screening.
* Subject accepting to keep the same lifestyle throughout the study regarding physical activity, no smoking etc.
* Registered with the French Social Security, in agreement with the French law on biomedical experimentation.

Exclusion Criteria:

* Subject with type 1 or 2 diabetes
* Smoker. Light smoker (less than 5 cigarettes per day) or former smoker (smoking more than 5 cigarettes per day) having stopped less than three months. Smoking (or use of smoking substitute e.g. nicotine patch) is not permitted from screening throughout the study.
* Subject with fasting capillary blood glucose level > 110 mg/dl.
* Subject with fasting capillary blood glucose level ≤ 110 mg/dl and 2 hours postprandial capillary blood glucose level > 140 mg/dl during an Oral Glucose Tolerance Test.
* Subject with any sensitivity or allergy to any of the products used within this clinical trial.
* Intake of product (food and dietary supplement) having an effect on glycemia and insulinemia.
* Intake of all chronic medication excepted oestroprogestative or progestative contraception started at least three months preceding the screening visit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Blood glucose incremental Area Under the Curve between 0 and 120 minutes after consumption of a standard meal, compared between MealShape and the placebo | Over 120 minutes after the consumption of a standard meal

SECONDARY OUTCOMES:
Blood glucose incremental Area Under the Curve between 0 and 60 minutes compared between MealShape and the placebo after consumption of a standard meal, | Over 60 minutes after consumption of a standard meal
Capillary blood glucose maximal concentration between MealShape and Placebo after consumption of a standard meal | Over 120 minutes after consumption of a standard meal
Comparison of glycemia values between MealShape and Placebo at the following time points: T0, T15, T30, T45, T60, T90 and T120 minutes after consumption of a standard meal | Over 120 minutes after consumption of a standard meal
Evaluation of the safety of MealShape with adverse events recording | 3 weeks
Insulin incremental Area under the Curve between 0 and 120 minutes compared between MealShape and Placebo after consumption of a standard meal | Over 120 minutes after consumption of a standard meal
Insulin incremental Area under the Curve between 0 and 60 minutes compared between MealShape and Placebo after consumption of a standard meal | Over 60 minutes after connsumption of a standard meal

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Deplanque, Principal Investigator — Naturalpha
Locations (1):
- Centre de Nutrition Clinique Naturalpha, Lilles, France

REFERENCES:
- [Background] Zimmet P, Alberti KG, Shaw J. Global and societal implications of the diabetes epidemic. Nature. 2001 Dec 13;414(6865):782-7. doi: 10.1038/414782a. PMID 11742409
- [Background] Finkelstein EA, Khavjou OA, Thompson H, Trogdon JG, Pan L, Sherry B, Dietz W. Obesity and severe obesity forecasts through 2030. Am J Prev Med. 2012 Jun;42(6):563-70. doi: 10.1016/j.amepre.2011.10.026. PMID 22608371
- [Background] Rafehi H, Ververis K, Karagiannis TC. Controversies surrounding the clinical potential of cinnamon for the management of diabetes. Diabetes Obes Metab. 2012 Jun;14(6):493-9. doi: 10.1111/j.1463-1326.2011.01538.x. Epub 2011 Dec 27. PMID 22093965
- [Background] Davis PA, Yokoyama W. Cinnamon intake lowers fasting blood glucose: meta-analysis. J Med Food. 2011 Sep;14(9):884-9. doi: 10.1089/jmf.2010.0180. Epub 2011 Apr 11. PMID 21480806
- [Background] Baker WL, Gutierrez-Williams G, White CM, Kluger J, Coleman CI. Effect of cinnamon on glucose control and lipid parameters. Diabetes Care. 2008 Jan;31(1):41-3. doi: 10.2337/dc07-1711. Epub 2007 Oct 1. PMID 17909085
- [Background] Magistrelli A, Chezem JC. Effect of ground cinnamon on postprandial blood glucose concentration in normal-weight and obese adults. J Acad Nutr Diet. 2012 Nov;112(11):1806-9. doi: 10.1016/j.jand.2012.07.037. PMID 23102179
- [Derived] Beejmohun V, Peytavy-Izard M, Mignon C, Muscente-Paque D, Deplanque X, Ripoll C, Chapal N. Acute effect of Ceylon cinnamon extract on postprandial glycemia: alpha-amylase inhibition, starch tolerance test in rats, and randomized crossover clinical trial in healthy volunteers. BMC Complement Altern Med. 2014 Sep 23;14:351. doi: 10.1186/1472-6882-14-351. PMID 25249234